CLINICAL TRIAL: NCT00967694
Title: Effect of N2O on Intraocular Pressure in Healthy Volunteers
Brief Title: Effect of Nitrous Oxide (N2O) on Intraocular Pressure in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Robert L. Bacon Medical Foundation (Unknown); Research to Prevent Blindness (Other)
Responsible Party: Principal Investigator, Kirk Lalwani, Associate Professor, Anesthesiology and Pediatrics, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00005402
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Glaucoma; Sedation
Keywords: Glaucoma; Nitrous oxide
MeSH Terms: conditions — Glaucoma | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitrous oxide administration (Experimental): All 20 healthy volunteers had their intraocular pressure (IOP) measured at baseline and then after 3, 6, 9, and 12 minutes of nitrous oxide administration, and then after 5, 10, and 15 minutes of breathing room air. There was therefore only one study arm, with each individual serving as their control for baseline and then intervention values of IOP measurement.
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — Nitrous oxide sedation by inhalation
  Other Names: N2O

SUMMARY:
The purpose of this study is to learn if breathing nitrous oxide (also known as "laughing gas") changes the pressure in a person's eyes. Some patients who need regular eye exams to measure their eye pressure often need to be put to sleep with medicine in order to complete the eye exam. Some of these medicines are known to cause changes in a person's eye pressure. Because of this, such medicines are avoided if the eye doctor needs to measure the patient's eye pressure. One medicine that is frequently used to put patients to sleep is nitrous oxide. No one really knows what effect nitrous oxide might have on a persons' eye pressure. The investigators are interested to see if nitrous oxide causes an increase, decrease, or no change in eye pressure. The investigators also want to investigate if there is a difference in the effects of nitrous oxide on eye pressure between males and females. Understanding these effects of nitrous oxide is important because during such eye exams, the eye doctor uses the pressure measurements to make important decisions about treatment and surgery options for the patient.

The investigators hypothesize that the use of inhaled nitrous oxide (N2O) will result in a decrease in IOP in healthy volunteers.

The investigators aim to determine the magnitude and duration of change, if any, in IOP caused by inhalation of N2O, and to assess if the gender of the patient has a role in this effect.

DETAILED DESCRIPTION:
An initial pre-anesthetic evaluation and physical examination will be performed by an attending anesthesiologist, and an eye exam will be performed by an attending ophthalmologist to determine suitability for inclusion according to the above criteria. Ideally the eye exam will take place immediately prior to conduction of the study. However, logistical restraints may require that the eye exam take place at a separate time/date prior to conduction of the study. IOPs will be measured by the attending ophthalmologist (B.E.) who will be blinded to the actual readings of the Tonopen by means of a small screen, and a single trained observer (E.F.) will record observations from the Tonopen. The nitrous oxide sedation will be managed by the attending anesthesiologist (K.L.). All patients will be monitored throughout using standardized monitoring (continuous EKG, non-invasive BP, and continuous pulse oximetry).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40
* American Society of Anesthesiologists Physical Classification System (ASA) Status 1-2
* Nil per os (NPO) prior to study (2 hrs clear liquids, 4 hrs milk, 6 hrs light food, 8 hrs heavy/greasy food)

Exclusion Criteria:

* Lack of volunteer consent
* Pregnancy
* History of features suggestive of a difficult airway on pre-anesthetic evaluation and physical examination
* Active gastroesophageal reflux disease
* Active obstructive sleep apnea
* History of recent trauma
* History of pneumothorax or lung cyst
* History of Vitamin B12 deficiency
* History of recent middle ear surgery (<3months)
* Current or recent (<3 weeks) respiratory tract infection
* Any acute illness or exacerbation of chronic illness such as asthma, chronic lung disease etc.
* Any history of cardiac ischemia (angina), myocardial infarction, or cardiac dysrhythmia.
* Myopia greater than -3 spherical equivalents or hyperopia greater than +3 spherical equivalents
* History of eye surgery of any sort, including refractive surgery, cataracts, and vitrectomy
* History of any ocular disease or infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Lalwani, MD,FRCA,MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrous Oxide Administration
Started | 26
Completed | 20 (5 discontinued during N2O administration due to agitation ⁄ dysphoria, one due to nausea⁄vomiting.)
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Volunteers recruited via locally placed posters, research opportunities website and email servers. Power calculations estimated 20 subjects would be needed to detect a 2.8mmHg difference in IOP. 26 subjects began nitrous oxide administration, with 6 choosing to withdraw. Baseline analysis based on the 20 participants completing the study.
Arm/Group | Nitrous Oxide Administration
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 26
American Society of Anesthesiologists Physical Classification System (ASA) class [Mean (Standard Deviation); unit: units on a scale] — Scale Range 1 to 6 with one being better, 6 being worst.
  ASA Physical Status 1 - A normal healthy patient ASA Physical Status 2 - A patient with mild systemic disease ASA Physical Status 3 - A patient with severe systemic disease ASA Physical Status 4 - A patient with severe systemic disease that is a constant threat to life ASA Physical Status 5 - A moribund patient who is not expected to survive without the operation ASA Physical Status 6 - A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 1.1 (0.307)
Baseline Mean Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHg] | 11.0 (2.4)
Baseline Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 86.4 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure During Nitrous Oxide Sedation
Time Frame: Before, during and after administration of nitrous oxide (45 minutes total)
Measure: Mean (95% Confidence Interval); unit: mmHg (difference in IOP)
Groups:
- Nitrous Oxide Administration: All 20 healthy volunteers had their intraocular pressure (IOP) measured at baseline (prior to nitrous oxide administration) and then after 3, 6, 9, and 12 minutes of nitrous oxide administration, and then after 5, 10, and 15 minutes of breathing room air. There was therefore one study arm, with each individual serving as their control for baseline (before nitrous oxide administration) and then intervention values of IOP measurement (during nitrous oxide administration), and then washout values of IOP (after breathing room air).
Arm/Group | Nitrous Oxide Administration
Number analyzed (Participants) | 20
mmHg (difference in IOP) | 1.05 [-0.81 to 2.9]
Statistical Analysis 1: Comparison: Nitrous Oxide Administration; A linear mixed effects model was used to assess change in IOP over time using time-points as the primary independent variable with significance set at p < 0.05. Power calculations showed that 20 subjects would allow detection of a 2.8-mmHg difference in IOP between any two time-points with 80% power assuming a standard deviation of 3.5 mmHg for IOP and a correlation between two time- points of 0.25; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Nitrous Oxide Administration: 20 healthy volunteers had their intraocular pressure (IOP) measured at baseline and then after 3, 6, 9, and 12 minutes of nitrous oxide administration, and then after 5, 10, and 15 minutes of breathing room air. There was therefore only one study arm, with each individual serving as their control for baseline and then intervention values of IOP measurement.
Arm/Group | Nitrous Oxide Administration
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 6/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide Administration (N=26)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) — 1 participants experienced transient, self-limited, mild nausea/vomiting and chose to withdraw from the study.
Dysphoria (Nervous system disorders) | 5 (5) — 5 participants experienced transient, self-limited, mild dysphoria and chose to withdraw from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No